CLINICAL TRIAL: NCT05722301
Title: Does Testosterone Therapy Improve Patient-Reported Outcomes in Age-Related Testosterone Deficient Patients Undergoing Total Hip Replacement: A Randomized-Controlled Trial
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: American Hip Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2019-08-16; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone Therapy (Experimental)
  Interventions: Drug: Testosterone Therapy
- No Testosterone Therapy (Placebo Comparator)
  Interventions: Other: No Testosterone Therapy

INTERVENTIONS:
Drug: Testosterone Therapy — The testosterone pellet implantation will be performed 2 weeks before surgery. The dose is determined by baseline levels of sex hormone binding globulin (SHBG) in the following manner: If SHBG > 60nmol/L implant 5 Testosterone Compounded 200mg (total 1000mgs testosterone). If SHBG 41-59 nmol/L implant 4 Testosterone Compounded 200mg (total 800mgs testosterone). If SHBG <40 nmol/L implant 3 Testosterone Compounded 200mg (total 600mgs testosterone).
  Arms: Testosterone Therapy
Other: No Testosterone Therapy — For the sham procedure no pellets will be implanted.
  Arms: No Testosterone Therapy

SUMMARY:
This randomized-controlled trial will study on the effect of testosterone therapy on patients undergoing total hip replacement. Subjects will be male patients > 50 years with testosterone deficiency undergoing total hip replacement due to severe degenerative joint disease. All participants will receive a total hip replacement and will be randomized to either testosterone therapy or placebo. A total of 80 subjects will be recruited randomized into 2 groups of 40 subjects. Testosterone therapy will be administered once to each patient at 2 weeks before surgery. The long-term follow up will be the same as all patients with patient-reported outcomes after total hip replacement, VAS for pain and satisfaction at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* 50 years of age and older
* Individuals who have degenerative joint disease requiring total hip replacement after failure of conservative measures.

Exclusion Criteria:

* History of prostate cancer less than 5 years ago or those men whom are not considered to be cancer free
* History of breast cancer less than 5 years ago or those men whom are not considered to be cancer free
* History of deep vein thrombosis (DVT)
* Presence of Factor V Leiden (as seen in labs)
* Presence of Protein S Deficiency (as seen in labs)
* History of atherosclerotic artery disease - by history having had a diagnosis made of CAD, MI, or stroke
* Liver disease (as viewed by liver function tests)
* Testosterone free level greater than 10pg/mL
* Hematocrit >51%; PSA >= 3ng/mL.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 3 months
  patient-reported outcome measure
Harris Hip Score | 1 year
  patient-reported outcome measure
Forgotten Joint Score | 3 months
  patient-reported outcome measure
Forgotten Joint Score | 1 year
  patient-reported outcome measure

SECONDARY OUTCOMES:
Visual Analog Scale | 3 months
  patient-reported outcome measure
Visual Analog Scale | 1 year
  patient-reported outcome measure
Patient Satisfaction (reported from questionnaire) | 3 months
  patient-reported outcome measure
Patient Satisfaction (reported from questionnaire) | 1 year
  patient-reported outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- American Hip Institute Research Foundation, Des Plaines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No